CLINICAL TRIAL: NCT02436356
Title: New Tools for Assessing Fracture Risk
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: FDA determined study device is significant risk. Study will not seek IDE.
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: ActiveLife Scientific (Industry); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Jeffry Nyman, Assistant Professor of Orthopaedics and Rehabilitation, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 141125; UL1TR000445 (NIH)
Record Dates: First submitted 2015-04-24; First posted 2015-05-06 (Estimated); Results first posted 2020-10-12 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Osteoporosis; Fracture Risk Assessment
MeSH Terms: conditions — Osteoporosis | interventions — Absorptiometry, Photon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Distal Radius Fracture Operative Group (Active Comparator): Fracture group patients will undergo DXA and MRI scans, along with Osteoprobe indentation.
  Interventions: Device: Osteoprobe-Reference Point Indentation (RPI); Radiation: Dual-energy X-ray absorptiometry (DXA) Scans; Radiation: MRI
- Healthy Volunteers (Non Fracture Group) (Active Comparator): Healthy volunteers will undergo DXA and MRI scans.
  Interventions: Radiation: Dual-energy X-ray absorptiometry (DXA) Scans; Radiation: MRI
- Distal Radius Fracture Non-operative Group (Active Comparator): Fracture group patients will undergo DXA and MRI scans, but will not undergo Osteoprobe indentation.
  Interventions: Radiation: Dual-energy X-ray absorptiometry (DXA) Scans; Radiation: MRI

INTERVENTIONS:
Device: Osteoprobe-Reference Point Indentation (RPI) — Diagnostic tool used for bone indentation to measure the ability of the tissue to resist microindentation (bone mineral strength).
  Arms: Distal Radius Fracture Operative Group
Radiation: Dual-energy X-ray absorptiometry (DXA) Scans — Assessment of Fracture Risk
Radiation: MRI — Determines bound water and pore water of bone.

SUMMARY:
The goal of this study is to determine whether two new, non-X-ray techniques can discriminate between high-energy fractures of normal bone (trauma) and low-energy fractures (fragility) of osteoporotic bone. The current gold-standard for assessing fracture risk areal bone mineral density (aBMD) by dual energy X-ray absorptiometry (DXA) is not particularly effective at identifying individuals who are at risk of suffering a fracture. Yet, there is a growing population of diabetics and elderly individuals prone to fractures. In effect, the age-related and diabetes-related increase in fracture risk is independent of a person's aBMD. These findings stress the urgency in developing diagnostic tools that can improve fracture risk prediction so that patients can be treated with the appropriate anti-fracture therapies.

ELIGIBILITY:
Inclusion/exclusion criteria for patients with a high-energy or fragility fracture requiring operative fixation (Arm 1)

Number of patients in Arm#1= 60 patients

Inclusion criteria:

1. Patients who are 18 years of age or older. This age range accounts for 60% of all distal radius fractures seen at Vanderbilt University Medical Center.
2. Patients who have sustained a low or high energy distal radius fracture that involves the metaphysis and requires open reduction internal fixation using volar plating.
3. English speaking due to feasibility of employing study personnel to deliver and assess study intervention.

Exclusion criteria:

1. Patients who have known risk factors of pathologic fractures (e.g. bone metastasis)
2. Patients who have or are receiving treatment for osteoporosis (e.g. bisphosphonate) lasted longer than 5 years
3. Patients who have Type 1 diabetes
4. Patients who have other bone disease (e.g., osteogenesis imperfecta, Paget's disease, thyroid disease, Vitamin D deficiency, hyperparathyroidism)
5. Patients that have a history of cancer, abnormal serum calcium, or chronic steroid use
6. Patients that would not be able to have a DXA scan (weight >350lbs, hardware in hips, patients that have lap band device)
7. Patients who are pregnant or who think they may be pregnant
8. Patients that have a medical contraindication to MRI (if patients are undergoing a study MRI)
9. Patients who have concurrent, bilateral upper extremity fractures where hardware or casting may affect study scan measurements
10. Patients who have distal radial shaft fractures

Exclusion criteria 1-5 are included because the goal of the study is to demonstrate whether new bone measurements differentiate normal bone from fragile bone. These exclusion criteria eliminate confounding factors that affect fracture resistance of bone in ways that are independent of osteoporosis. Exclusion criteria 6-8 are practical since DXA/MRI scans cannot accommodate all people.

Inclusion/exclusion criteria for patients with no fracture (Arm 2)

Number of patients in Arm#2= 40 patients

Inclusion criteria:

1. Patients who are 18 years of age or older.
2. Patients who have no history of fracture or family history of pathologic fracture
3. English speaking due to feasibility of employing study personnel to deliver and assess study intervention.

Exclusion criteria:

1. Patients who are taking medication to treat osteoporosis (e.g. bisphosphonate)
2. Patients who have or are receiving treatment for osteoporosis (e.g. bisphosphonate) lasted longer than 5 years
3. Patients who have Type 1 diabetes
4. Patients who have other bone disease (e.g., osteogenesis imperfecta, Paget's disease, thyroid disease, Vitamin D deficiency, hyperparathyroidism).
5. Patients that have a history of cancer, abnormal serum calcium, or chronic steroid use.
6. Patients that would not be able to have a DXA scan (weight >350lbs, hardware in hips, patients that have lap band device)
7. Patients who are pregnant or who think they may be pregnant.
8. Patients that have a medical contraindication to MRI.

Exclusion criteria 1-5 are included because the goal of the study is to demonstrate whether new bone measurements differentiate normal bone from fragile bone. These exclusion criteria eliminate confounding factors that affect fracture resistance of bone in ways that are independent of osteoporosis. Exclusion criteria 6- 8 are practical since DXA/MRI scans cannot accommodate all people.

Inclusion/exclusion criteria for patients with a high-energy or fragility fracture requiring nonoperative treatment (Arm 3)

Number of patients in Arm#3= up to 10 patients

Inclusion criteria:

1. Patients who are 18 years of age or older. This age range accounts for 60% of all distal radius fractures seen at Vanderbilt University Medical Center.
2. Patients who have sustained a low or high energy distal radius fracture that requires nonoperative treatment
3. English speaking due to feasibility of employing study personnel to deliver and assess study intervention.

Exclusion criteria:

1. Patients who have known risk factors of pathologic fractures (e.g. bone metastasis)
2. Patients who have or are receiving treatment for osteoporosis (e.g. bisphosphonate) lasted longer than 5 years
3. Patients who have Type 1 diabetes
4. Patients who have other bone disease (e.g., osteogenesis imperfecta, Paget's disease, thyroid disease, Vitamin D deficiency, hyperparathyroidism)
5. Patients that have a history of cancer, abnormal serum calcium, or chronic steroid use
6. Patients that would not be able to have a DXA scan (weight >350lbs, hardware in hips, patients that have lap band device)
7. Patients who are pregnant or who think they may be pregnant
8. Patients that have a medical contraindication to MRI (if patients are undergoing a study MRI)
9. Patients who have concurrent, bilateral upper extremity fractures where hardware or casting may affect study scan measurements

Exclusion criteria 1-5 are included because the goal of the study is to demonstrate whether new bone measurements differentiate normal bone from fragile bone. These exclusion criteria eliminate confounding factors that affect fracture resistance of bone in ways that are independent of osteoporosis. Exclusion criteria 6-8 are practical since DXA/MRI scans cannot accommodate all people.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-06-30 (Actual); Primary Completion 2018-05-23 (Actual); Study Completion 2018-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffry S Nyman, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Univeristy Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
No current plant to share individual participant data.

RESULTS

PARTICIPANT FLOW:
Groups:
- Distal Radius Fracture Operative Group: Fracture group patients will undergo DXA and MRI scans, along with Osteoprobe indentation.
  Osteoprobe-RPI (Reference Point Indentation): Diagnostic tool used for bone indentation to measure the ability of the tissue to resist microindentation (bone mineral strength).
  Dual-energy X-ray absorptiometry (DXA) Scans: Assessment of Fracture Risk
  MRI: Determines bound water and pore water of bone.
Period: Overall Study
Arm/Group | Distal Radius Fracture Operative Group | Healthy Volunteers (Non Fracture Group) | Distal Radius Fracture Non-operative Group
Started | 33 | 11 | 4
High Energy Fracture | 14 | 0 | 4
Low Energy Fracture | 19 | 0 | 0
Completed | 28 | 10 | 2
Not Completed | 5 | 1 | 2
Not completed — Excluded by MRI Screening | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Surgical Approach (Dorsal not volar) | 1 | 0 | 0
Not completed — Excluded due to other medical conditions | 3 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline Characteristics section does not include demographics data of 5 Distal Radius Operative Arm subjects, 1 Healthy Volunteer Arm subject and 2 Distal Radius Nonoperative Arm subjects. These subjects were withdrawn/lost to follow-up following consent, but prior to any study procedures taking place.
Groups:
- Distal Radius Fracture Operative Group: Fracture group patients will undergo DXA and MRI scans, along with Osteoprobe indentation.
  Osteoprobe-RPI: Diagnostic tool used for bone indentation to measure the ability of the tissue to resist microindentation (bone mineral strength).
  Dual-energy X-ray absorptiometry (DXA) Scans: Assessment of Fracture Risk
  MRI: Determines bound water and pore water of bone.
- Total: Total of all reporting groups
Arm/Group | Distal Radius Fracture Operative Group | Healthy Volunteers (Non Fracture Group) | Distal Radius Fracture Non-operative Group | Total
Number analyzed (Participants) | 28 | 10 | 2 | 40
Age, Continuous [Mean (Full Range); unit: years] | 47 [18 to 76] | 44 [24 to 63] | 30 [25 to 35] | 40 [18 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 7 | 0 | 26
  Male | 9 | 3 | 2 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 26 | 9 | 2 | 37
  Unknown or Not Reported | 2 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 0 | 3
  White | 25 | 10 | 2 | 37
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 10 | 2 | 40
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m2] — Population: BMI unavailable for one subject in distal radius fracture operative group.
  kg/m2
    number analyzed (Participants) | 27 | 10 | 2 | 39
    (all) | 27.9 [17.2 to 41.5] | 27.55 [18.16 to 39.34] | 25.61 [22.07 to 29.16] | 27.7 [17.2 to 41.5]

OUTCOME MEASURES:

1. Primary Outcome: Osteoprobe Measurements
Description: Bone Material Strength index (BMSi)
  By engaging the bone at 10 N and then delivering a single impact force of ~40 N, the OsteoProbe records the maximum penetration depth of conical-spherical tip into cortical bone. This indentation distance increase (IDI) is indexed to the IDI acquired from a reference material immediately after the bone IDI measurements, such that the OsteoProbe-based measurement known as bone material strength index (BMSi) is 100 times IDI of reference material divided by IDI of the patient's bone. A lower BMSi measurement is the result of a higher indentation distance into the bone. For statistical analysis, we used the mean of the 10 BMSi measurements per case.
Time Frame: Within a week before or after surgery to repair distal radius fracture
Population: Only Distal Radius Fracture Operative Group subjects underwent Osteoprobe measurements where Bone Material Strength index (BMSi) was obtained.
Measure: Median (95% Confidence Interval); unit: Index
Groups:
- Distal Radius Fracture Operative Group: Distal Radius Fracture Operative group patients will undergo DXA and MRI scans, along with Osteoprobe indentation.
  Osteoprobe-RPI: Diagnostic tool used for bone indentation to measure the ability of the tissue to resist microindentation (bone mineral strength).
  Dual-energy X-ray absorptiometry (DXA) Scans: Assessment of Fracture Risk
  MRI: Determines bound water and pore water of bone.
- Healthy Volunteers: Healthy volunteers will undergo DXA and MRI scans.
  Dual-energy X-ray absorptiometry (DXA) Scans: Assessment of Fracture Risk
  MRI: Determines bound water and pore water of bone.
- Distal Radius Fracture Non-Operative Group: Distal Radius Fracture Non-Operative group patients will undergo DXA and MRI scans.
  Dual-energy X-ray absorptiometry (DXA) Scans: Assessment of Fracture Risk
  MRI: Determines bound water and pore water of bone.
Arm/Group | Distal Radius Fracture Operative Group | Healthy Volunteers | Distal Radius Fracture Non-Operative Group
Number analyzed (Participants) | 28 | 0 | 0
Index
  High Energy: number analyzed (Participants) | 11 | 0 | 0
  High Energy | 73.3 [60.2 to 79.8] |  |
  Low Energy: number analyzed (Participants) | 17 | 0 | 0
  Low Energy | 76.3 [70.1 to 79] |  |

2. Primary Outcome: MRI Scan Measurements
Description: Bound Water Fraction
Time Frame: Within a week before or after surgery to repair distal radius fracture
Population: Distal Radius Fracture Nonoperative Group- 2 subjects did not have MRI scan data.
  Healthy Volunteers- 1 subject did not take part in the MRI scan.
  Distal Radius Fracture Operative Group- 8 Low Energy and 6 high energy subjects did not take part in the MRI scan. 3 high energy subjects did not have usable MRI data due to technical issues.
Measure: Median (95% Confidence Interval); unit: percentage of bound water fraction
Groups:
- Distal Radius Fracture Operative Group: Distal Radius Fracture Operative Group subjects will undergo DXA and MRI scans, along with Osteoprobe indentation.
  Osteoprobe-RPI: Diagnostic tool used for bone indentation to measure the ability of the tissue to resist microindentation (bone mineral strength).
  Dual-energy X-ray absorptiometry (DXA) Scans: Assessment of Fracture Risk
  MRI: Determines bound water and pore water of bone.
- Distal Radius Fracture Non-operative Group: Distal Radius Fracture Non-operative Group subjects will undergo DXA and MRI scans.
  Dual-energy X-ray absorptiometry (DXA) Scans: Assessment of Fracture Risk
  MRI: Determines bound water and pore water of bone.
Arm/Group | Distal Radius Fracture Operative Group | Healthy Volunteers | Distal Radius Fracture Non-operative Group
Number analyzed (Participants) | 14 | 10 | 0
percentage of bound water fraction
  High Energy Fracture: number analyzed (Participants) | 5 | 0 | 0
  High Energy Fracture | 12.6 [9.51 to 33] |  |
  Low Energy Fracture: number analyzed (Participants) | 14 | 0 | 0
  Low Energy Fracture | 16.6 [12.8 to 20.0] |  |
  No fracture: number analyzed (Participants) | 0 | 10 | 0
  No fracture |  | 25.9 [21.1 to 30.2] |

3. Primary Outcome: MRI Scan Measurements
Description: Pore Water Fraction
Time Frame: Within a week before or after surgery to repair distal radius fracture
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: percentage of pore water fraction
Arm/Group | Distal Radius Fracture Operative Group | Healthy Volunteers | Distal Radius Fracture Non-operative Group
Number analyzed (Participants) | 14 | 10 | 0
percentage of pore water fraction
  High Energy Fracture: number analyzed (Participants) | 5 | 0 | 0
  High Energy Fracture | 12.9 [1.86 to 17.1] |  |
  Low Energy Fracture: number analyzed (Participants) | 14 | 0 | 0
  Low Energy Fracture | 17.4 [8.5 to 22.7] |  |
  No fracture: number analyzed (Participants) | 0 | 10 | 0
  No fracture |  | 10.4 [7.7 to 12.1] |

4. Primary Outcome: DXA Scan Measurements
Description: Bone Mineral Density
Time Frame: Within a week before or after surgery to repair distal radius fracture
Population: Distal Radius Fracture Operative Group- Includes 9 high energy fracture and 14 low energy fracture subjects.
  High Energy: 1 did not have L1-L4 scanned, 2 did not receive calculations due to age. Low Energy- 3 did not have a DXA scan.
  Healthy Volunteers- 1 subject did not have a DXA scan.
Measure: Median (95% Confidence Interval); unit: g/cm^2
Arm/Group | Distal Radius Fracture Operative Group | Healthy Volunteers | Distal Radius Fracture Non-operative Group
Number analyzed (Participants) | 23 | 10 | 2
g/cm^2
  High Energy- L1 -L4 VB: number analyzed (Participants) | 8 | 0 | 2
  High Energy- L1 -L4 VB | 1.119 [1.022 to 1.546] |  | 1.475 [1.022 to 1.475]
  Low Energy- L1-L4 VB: number analyzed (Participants) | 14 | 0 | 0
  Low Energy- L1-L4 VB | 1.165 [1.058 to 1.322] |  |
  No Fracture- L1-L4 VB: number analyzed (Participants) | 0 | 10 | 0
  No Fracture- L1-L4 VB |  | 1.138 [0.908 to 1.302] |
  High Energy- Hip: number analyzed (Participants) | 9 | 0 | 2
  High Energy- Hip | 1.088 [0.949 to 1.213] |  | 1.197 [0.902 to 1.197]
  Low Energy- Hip: number analyzed (Participants) | 14 | 0 | 0
  Low Energy- Hip | 0.909 [0.798 to 1.024] |  |
  No Fracture- Hip: number analyzed (Participants) | 0 | 10 | 0
  No Fracture- Hip |  | 0.988 [0.777 to 1.140] |
  High Energy- Femur neck: number analyzed (Participants) | 9 | 0 | 2
  High Energy- Femur neck | 1.063 [0.876 to 1.167] |  | 1.322 [0.849 to 1.322]
  Low Energy- Femur neck: number analyzed (Participants) | 14 | 0 | 0
  Low Energy- Femur neck | 0.920 [0.825 to 1.039] |  |
  No fracture- Femur neck: number analyzed (Participants) | 0 | 10 | 0
  No fracture- Femur neck |  | 1.008 [0.753 to 1.135] |
  High Energy- Radius distal-third: number analyzed (Participants) | 9 | 0 | 2
  High Energy- Radius distal-third | 0.938 [0.754 to 1.041] |  | 1.059 [0.851 to 1.059]
  Low Energy- Radius distal-third: number analyzed (Participants) | 14 | 0 | 0
  Low Energy- Radius distal-third | 0.833 [0.695 to 0.958] |  |
  No Fracture- Radius distal-third: number analyzed (Participants) | 0 | 10 | 0
  No Fracture- Radius distal-third |  | 0.887 [0.683 to 1.069] |
  High Energy- Radius ultra-distal: number analyzed (Participants) | 9 | 0 | 2
  High Energy- Radius ultra-distal | 0.924 [0.743 to 1.128] |  | 1.071 [0.837 to 1.071]
  Low Energy- Radius ultra-distal: number analyzed (Participants) | 14 | 0 | 0
  Low Energy- Radius ultra-distal | 0.810 [0.647 to 0.908] |  |
  No Fracture- Radius ultra-distal: number analyzed (Participants) | 0 | 10 | 0
  No Fracture- Radius ultra-distal |  | 0.883 [0.761 to 1.043] |

5. Primary Outcome: DXA Scan Measurements
Description: Bone Mineral Content
Time Frame: Within a week before or after surgery to repair distal radius fracture
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: g
Arm/Group | Distal Radius Fracture Operative Group | Healthy Volunteers | Distal Radius Fracture Non-operative Group
Number analyzed (Participants) | 23 | 10 | 2
g
  High Energy L1-L4 VB: number analyzed (Participants) | 8 | 0 | 2
  High Energy L1-L4 VB | 65.04 [50.54 to 101.70] |  | 98.87 [58.63 to 98.87]
  Low Energy L1-L4 VB: number analyzed (Participants) | 14 | 0 | 0
  Low Energy L1-L4 VB | 74.24 [53.21 to 74.61] |  |
  No Fracture L1-L4 VB: number analyzed (Participants) | 0 | 10 | 0
  No Fracture L1-L4 VB |  | 70.19 [47.86 to 74.91] |
  High Energy- Hip: number analyzed (Participants) | 9 | 0 | 2
  High Energy- Hip | 43.03 [29.37 to 47.17] |  | 44.97 [31.56 to 44.97]
  Low Energy- Hip: number analyzed (Participants) | 14 | 0 | 0
  Low Energy- Hip | 33.5 [25.6 to 35.88] |  |
  No Fracture- Hip: number analyzed (Participants) | 0 | 10 | 0
  No Fracture- Hip |  | 36.97 [22.43 to 38.38] |
  High Energy- Femur neck: number analyzed (Participants) | 9 | 0 | 2
  High Energy- Femur neck | 6.05 [4.32 to 6.30] |  | 7.26 [4.58 to 7.26]
  Low Energy- Femur neck: number analyzed (Participants) | 14 | 0 | 0
  Low Energy- Femur neck | 4.848 [3.99 to 5.05] |  |
  No Fracture- Femur neck: number analyzed (Participants) | 0 | 10 | 0
  No Fracture- Femur neck |  | 5.49 [3.73 to 6.11] |
  High Energy- Radius distal-third: number analyzed (Participants) | 9 | 0 | 2
  High Energy- Radius distal-third | 3.07 [1.76 to 3.38] |  | 3.64 [2.09 to 3.64]
  Low Energy- Radius distal-third: number analyzed (Participants) | 14 | 0 | 0
  Low Energy- Radius distal-third | 2.433 [1.7 to 2.59] |  |
  No Fracture- Radius distal-third: number analyzed (Participants) | 0 | 10 | 0
  No Fracture- Radius distal-third |  | 2.43 [1.84 to 2.57] |
  High Energy- Radius ultra-distal: number analyzed (Participants) | 9 | 0 | 2
  High Energy- Radius ultra-distal | 2.39 [1.35 to 2.67] |  | 2.43 [1.64 to 2.43]
  Low Energy- Radius ultra-distal: number analyzed (Participants) | 14 | 0 | 0
  Low Energy- Radius ultra-distal | 1.713 [1.03 to 1.96] |  |
  No Fracture- Radius ultra-distal: number analyzed (Participants) | 0 | 10 | 0
  No Fracture- Radius ultra-distal |  | 1.87 [1.23 to 2.04] |

6. Primary Outcome: DXA Scan Measurements
Description: A T-score is the number of standard deviations (SD) below (negative value) or above (positive value) the mean BMD (bone mineral density) for a healthy population. A person with T-score below -2.5 is considered to have osteoporosis.
Time Frame: Within a week before or after surgery to repair distal radius fracture
Population: Distal Radius Fracture Operative Group- Includes 7 high energy fracture and 14 low energy fracture subjects.
  High Energy: 1 did not have L1-L4 scanned, 2 did not receive calculations due to age. Low Energy- 3 did not have a DXA scan.
  Healthy Volunteers- 1 subject did not have a DXA scan.
Measure: Median (95% Confidence Interval); unit: t-score
Arm/Group | Distal Radius Fracture Operative Group | Healthy Volunteers | Distal Radius Fracture Non-operative Group
Number analyzed (Participants) | 21 | 10 | 2
t-score
  High Energy- L1-L4 VB: number analyzed (Participants) | 6 | 0 | 2
  High Energy- L1-L4 VB | 0.8 [-1.3 to 2.5] |  | 1.9 [-1.7 to 1.9]
  Low Energy- L1-L4 VB: number analyzed (Participants) | 14 | 0 | 0
  Low Energy- L1-L4 VB | 0.6 [-1.5 to 0.7] |  |
  No Fracture- L1-L4 VB: number analyzed (Participants) | 0 | 10 | 0
  No Fracture- L1-L4 VB |  | 0.5 [-2.3 to 0.6] |
  High Energy- Hip: number analyzed (Participants) | 7 | 0 | 2
  High Energy- Hip | 1.2 [-1.7 to 1.6] |  | 0.8 [-1.4 to 0.8]
  Low Energy- Hip: number analyzed (Participants) | 14 | 0 | 0
  Low Energy- Hip | -0.2 [-1.7 to -0.1] |  |
  No Fracture- Hip: number analyzed (Participants) | 0 | 10 | 0
  No Fracture- Hip |  | 0.7 [-1.8 to 0.8] |
  High Energy- Femur neck: number analyzed (Participants) | 7 | 0 | 2
  High Energy- Femur neck | 0.7 [-1.3 to 1.4] |  | 1.9 [-1.7 to 1.9]
  Low Energy- Femur neck: number analyzed (Participants) | 14 | 0 | 0
  Low Energy- Femur neck | -0.4 [-1.5 to -0.2] |  |
  No Fracture- Femur neck: number analyzed (Participants) | 0 | 10 | 0
  No Fracture- Femur neck |  | 0.3 [-2.1 to 0.5] |
  High Energy- Radius distal-third: number analyzed (Participants) | 7 | 0 | 2
  High Energy- Radius distal-third | 0.7 [-2.2 to 0.7] |  | 0.7 [-1.4 to 0.7]
  Low Energy- Radius distal-third: number analyzed (Participants) | 14 | 0 | 0
  Low Energy- Radius distal-third | 0.8 [-2.1 to 0.9] |  |
  No Fracture- Radius distal-third: number analyzed (Participants) | 0 | 10 | 0
  No Fracture- Radius distal-third |  | 0.6 [-2.2 to 0.8] |
  High Energy- Radius ultra-distal: number analyzed (Participants) | 7 | 0 | 2
  High Energy- Radius ultra-distal | 1.3 [-4.0 to 3.9] |  | 1.3 [-2.3 to 1.3]
  Low Energy- Radius ultra-distal: number analyzed (Participants) | 14 | 0 | 0
  Low Energy- Radius ultra-distal | -1.0 [-4.2 to -0.2] |  |
  No Fracture- Radius ultra-distal: number analyzed (Participants) | 0 | 10 | 0
  No Fracture- Radius ultra-distal |  | 0.2 [-0.8 to 0.4] |

7. Secondary Outcome: Patient-reported Measurements
Description: DASH (Disabilities of the Arm, Shoulder, and Hand) is a 30-item self-report questionnaire designed to assess musculoskeletal disorders of the upper limbs. The score ranges from 0 (no disability) to 100 (most severe disability). A higher scores indicate a greater level of disability and severity, whereas, lower scores indicate a lower level of disability.
Time Frame: Baseline/One-Time Completion and Post-op/-treatment: 3, 6, and 12 weeks
Population: Distal Radius Fracture Operative Group- Includes 11 high energy fracture and 17 low energy fracture subjects.
  Healthy Volunteers were only asked to complete the DASH at the baseline visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Distal Radius Fracture Operative Group | Healthy Volunteers | Distal Radius Fracture Non-operative Group
Number analyzed (Participants) | 28 | 10 | 2
score on a scale
  High Energy- Baseline: number analyzed (Participants) | 11 | 0 | 2
  High Energy- Baseline | 41.18 (28.08) |  | 27.66 (6.83)
  Low Energy- Baseline: number analyzed (Participants) | 16 | 0 | 0
  Low Energy- Baseline | 59.89 (18.50) |  |
  No Fracture- Baseline: number analyzed (Participants) | 0 | 9 | 0
  No Fracture- Baseline |  | 0.83 (1.04) |
  High Energy- 3 Week: number analyzed (Participants) | 9 | 0 | 2
  High Energy- 3 Week | 35.39 (25.13) |  | 7.50 (6.66)
  Low Energy- 3 Week: number analyzed (Participants) | 14 | 0 | 0
  Low Energy- 3 Week | 50.73 (18.85) |  |
  High Energy- 6 Week: number analyzed (Participants) | 10 | 0 | 2
  High Energy- 6 Week | 28.43 (24.46) |  | 38.93 (20.98)
  Low Energy- 6 Week: number analyzed (Participants) | 28 | 0 | 0
  Low Energy- 6 Week | 38.93 (20.98) |  |
  High Energy- 12 Week: number analyzed (Participants) | 7 | 0 | 2
  High Energy- 12 Week | 3.33 (4.45) |  | 0.84 (0.84)
  Low Energy- 12 Week: number analyzed (Participants) | 15 | 0 | 0
  Low Energy- 12 Week | 21.92 (20.67) |  |

8. Secondary Outcome: Patient-reported Measurements
Description: PRWE (Patient-rated wrist evaluation) is a 15-item survey designed to measure wrist pain and disability in activities of daily living. The PRWE consists of a pain subscale and a function subscale. The pain subscale contains 5 items, each rated 0 (no pain) to 10 (worst pain ever). The pain subscale is calculated by adding all 5 item scores together (minimum score: 0, maximum score: 50). A lower score indicates a lower pain level. The function subscale contains 10 items, each rated 0 (no difficulty) to 10 (unable to do). The function subscale is calculated by adding all 10 item scores together and dividing by 2 (minimum score: 0, maximum score: 100). A lower score indicates a lower disability level. The total PRWE score is calculated by adding the pain and function subscales together. The total PRWE score ranges from 0 (best score) to 100 (worst score). The lower the score the better the outcome.
Time Frame: Baseline and Post-op/-treatment: 3, 6, and 12 weeks
Population: Only subjects with a fracture were asked to complete the PRWE survey. Distal Radius Fracture Operative Group- Includes 11 high energy fracture and 17 low energy fracture subjects.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Distal Radius Fracture Operative Group | Healthy Volunteers | Distal Radius Fracture Non-operative Group
Number analyzed (Participants) | 28 | 0 | 2
score on a scale
  High Energy- Baseline: number analyzed (Participants) | 11 | 0 | 2
  High Energy- Baseline | 70.45 (18.89) |  | 43.5 (4.5)
  Low Energy- Baseline: number analyzed (Participants) | 17 | 0 | 0
  Low Energy- Baseline | 76.30 (16.85) |  |
  High Energy- 3 Week: number analyzed (Participants) | 9 | 0 | 2
  High Energy- 3 Week | 52.44 (27.04) |  | 13.5 (7.5)
  Low Energy- 3 Week: number analyzed (Participants) | 14 | 0 | 0
  Low Energy- 3 Week | 61.11 (15.29) |  |
  High Energy- 6 Week: number analyzed (Participants) | 10 | 0 | 2
  High Energy- 6 Week | 39.53 (24.89) |  | 10 (6)
  Low Energy- 6 Week: number analyzed (Participants) | 16 | 0 | 0
  Low Energy- 6 Week | 47.69 (25.43) |  |
  High Energy-12 Week: number analyzed (Participants) | 7 | 0 | 2
  High Energy-12 Week | 5.29 (5.37) |  | 2 (2)
  Low Energy- 12 Week: number analyzed (Participants) | 15 | 0 | 0
  Low Energy- 12 Week | 28.23 (25.99) |  |

ADVERSE EVENTS:
Time Frame: 12 weeks for distal radius fracture patients 0 weeks for healthy volunteers
Description: Non-serious Adverse Event- An infection or bleeding in a patient as a result of their distal radius fracture plating surgery with Osteoprobe use.
Arm/Group | Distal Radius Fracture Operative Group | Healthy Volunteers (Non Fracture Group) | Distal Radius Fracture Non-operative Group
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/10 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/10 | 0/2
Other Adverse Events (participants affected / at risk) | 0/28 | 0/10 | 0/2

LIMITATIONS AND CAVEATS:
Early termination of the study occurred in February 2020 when the FDA determined the OsteoProbe is a significant risk device that would require an IDE (Investigational Device Exemption).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has 30 days prior to proposed submission date/release of publication to review results, provide comments. Within 30 days of receipt of proposed publication, Sponsor shall advise PI in writing if information contains Sponsor's confidential information (CI) or patentable matter. In addition, upon written request by Sponsor, PI shall delay submission of such publication for an additional 60 days in order to allow Active Life to apply for patent or other protection for Sponsor inventions.

DOCUMENTS (3):
  • Study Protocol (2017-03-08): https://cdn.clinicaltrials.gov/large-docs/56/NCT02436356/Prot_001.pdf
  • Statistical Analysis Plan (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/56/NCT02436356/SAP_002.pdf
  • Informed Consent Form (2015-09-24): https://cdn.clinicaltrials.gov/large-docs/56/NCT02436356/ICF_003.pdf